CLINICAL TRIAL: NCT05343208
Title: Effectiveness of Online Therapy to Prevent Burnout
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: SciensCollege (Industry)
Collaborators: Karlstad University (Other); My-E-Health (Unknown)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: SC-EOTPB-1
Record Dates: First submitted 2022-04-14; First posted 2022-04-25 (Actual); Last update posted 2022-04-25 (Actual); Status verified 2022-04

CONDITIONS: Burnout; Risk Reduction; Cognitive Change
Keywords: Prevention; Mental Health; Cognitive Behavioral Therapy; Interactive Online Therapy; TeleHealth
MeSH Terms: conditions — Burnout, Psychological; Risk Reduction Behavior; Psychological Well-Being

STUDY DESIGN:
Intervention Model Description: An empirical and parallel design using raw EFP psychometric data to measure the effectiveness of online therapy to reduce the risk for Burnout between a control group and an online therapy group.
Masking Description: Randomly selected from an employer list
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Cognitive Behavioral Therapy Group (Experimental): The group received online Cognitive Behavioral Therapy via the My-E-Health. Patients were issued a preTest psychometric assessment and a post therapy assessment using the Burnout Psychometrics provided within the My-E-Health's online ecosystem. All patients were required to validate the accuracy of the assessments during a follow-up of their results.
  Interventions: Diagnostic Test: EFP Psychometric assessment to determine level of afflication
- Control Group (No Intervention): The Control Group received no online therapy. Patients were issued a preTest psychometric assessment and a post therapy assessment using the Burnout Psychometrics provided within the My-E-Health's online ecosystem. All patients were required to validate the accuracy of the assessments during a follow-up of their results.

INTERVENTIONS:
Diagnostic Test: EFP Psychometric assessment to determine level of afflication — Patients were asked to complete a psychometric assessment in relation to their psychological wellbeing. Results were presented to the patient and validdated by the patient.
  Arms: Cognitive Behavioral Therapy Group

SUMMARY:
This study aims to address the reliability and validity of the Empowerment for Participation (EFP) batch of assessments to measure Burnout risk in relation to the efficacy of online interventions to provide proactive rehabilitation using Cognitive Behavioral Therapy (CBT) and floating to achieve improved mental health and wellbeing.

DETAILED DESCRIPTION:
An Empirical design using raw EFP psychometric data to measure the effectiveness of online therapy to reduce the risk for Burnout between a control group and an online therapy group. The aim is to test whether or not there is a statistically significant difference in the effectiveness on online therapy to reduce the Risk for Burnout compared to that of a Control Group. Fifty participants were randomly selected. The rehabilitation and control Group consisted of twenty-five normally distributed employees (N25) each. The rehabilitation group received therapy, and the control had not yet received any form of therapy. SPSS was used to analyze the data collected, a Repeated Measure ANOVA, an ANCOVA, a Discriminant analysis, and a Construct Validity analysis were used to test for Reliability and Validity.

The group was randomly selected from a list of employees within the My-E-Health ecosystem. The group (N50) normally distributed group met all assumptions and consisted of a Control Group (N25) and a Therapy Group (N25). The post assessment value was used as the dependent variable.

The Burnout measure (30 questions) is obtained from the Empowerment for Participation (EFP) batch of assessments (110 questions). All assessments and CBT were done digitally online and floating was done at a designated location. The full EFP assessment is integrated into a digital ecosystem designed for this purpose and therapy. The online digital system is an integrity-based platform offering both the employee and caregiver a secure and encrypted ecosystem or secure data tunnel or channel between the therapists and patients.

ELIGIBILITY:
Inclusion Criteria

Employees assessed on the EFP Burnout Scale as having:

* a Moderate Risk of Burnout
* a High Risk of Burnout
* A Burned out Risk (Mental Health Exhaustion)
* Employees with a current Bunrout diagnosis from a hospital, outpatient or psychiatric cllinic
* A fully employed person with a member organization
* No other inclusion criteria.

Exclusion Criteria:

Employees assessed on the EFP Burnout Scale as having:

* No evidence of Burnout
* Low Risk of Burnout.
* Unemployed persons
* No other exclusion critera was used.

Ages: 22 Years to 68 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 1916-09-05 (Actual); Primary Completion 2021-01-11 (Actual); Study Completion 2022-04-04 (Actual)

PRIMARY OUTCOMES:
To measure the difference between a pre- and post-assessment score for Burnout in a Control Group versus a Therapy Group. | From admission to discharge, up to 3 months.
  The Burnout measure (30 questions) is obtained from the Empowerment for Participation (EFP) batch of assessments using Visual Analog Scales (VAS) online. A straight line with a beginning and end point. As the slider moves from left to right, the text positioned at either end of the line increases as the opposite end decreases. The position where the slider stops is represented by a number from 0-20.
  The risk assessment scale (0-600) determines the level of intervention and preventive care.
  There are five risk levels of Burnout in relation to the total score following a lineal guide: 0-99 points (M=0-3.300) = No evidence of Burnout, 100-199 points (M=3.333-6.6333) = Low risk for Burnout, 200-299 points (M=6.6667-9.9667) = Moderate risk for Burnout, 300-399 points (M=10.00-13.300) = High risk for Burnout, and 400-600 points (M=13.3333-20) = Burnout. Patient content validation and score accuracy is required after each assessment.

CONTACTS AND LOCATIONS:
Overall Officials: Clive S Michelsen, M.Sc., Principal Investigator — SciensCollege
Locations (1):
- SciensCollege, Malmo, Skåne County, Sweden

IPD SHARING:
Plan to Share IPD: Yes
All IPD that underlie results in a publication. SPSS files.
Supporting Information: SAP
Time Frame: The data is available from April 15, 2022 for one year until April 14th, 2023
Access Criteria: contact clive@scienscollege.se with your reason for this research and your contact details. You'll be forwarded the SPSS data file.

REFERENCES:
- [Derived] Michelsen C, Kjellgren A. The Effectiveness of Web-Based Psychotherapy to Treat and Prevent Burnout: Controlled Trial. JMIR Form Res. 2022 Aug 11;6(8):e39129. doi: 10.2196/39129. PMID 35802001